CLINICAL TRIAL: NCT07142759
Title: Investigating the Impact of Vitamin D Biofortified Tomatoes on Serum Levels of 25(OH)D - a Two Phase, a Randomized Double-blind Placebo-controlled Parallel Arm Trial (RCT)
Brief Title: Investigating the Impact of Vitamin D Biofortified Tomatoes on Serum Levels of 25(OH)D
Acronym: ViTaL-D
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: University of Surrey (Other); John Innes Centre (Unknown); Norfolk and Norwich University Hospitals NHS Foundation Trust (Other); NIHR Norfolk Clinical Research Facility (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: QIB03/2024; IRAS 349335 (Other: Health Research Authority)
Record Dates: First submitted 2025-08-19; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Vitamin D Insufficiency
Keywords: tomato soup; precision breeding; biofortification; vitamin D; 25-hydroxy vitamin D (25[OH]D); dietary intervention

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soup with Precision Bred Tomatoes (Provitamin D-rich, No UV-Treatment) (Experimental): Soup made with precision bred (gene-edited) tomatoes that have been engineered to accumulate 7-dehydrocholesterol (7-DHC) also known as provitamin D is a precursor of vitamin D3. These tomatoes have undergone CRISPR-Cas9 gene editing to allow the accumulation of 7-DHC in the tomatoes and remains to be rich in 7-DHC when protected from UV light.
  Interventions: Other: Precision Bred Provitamin D-rich Tomato Soup
- Soup with Precision Bred Tomatoes (Vitamin D-rich, UV-Treated) (Experimental): Soup is made with the same precision bred tomatoes, but in this case, the tomatoes have been treated with ultraviolet (UV) light to convert the accumulated 7-DHC into vitamin D3. UV exposure mimics the natural process by which human skin synthesizes vitamin D3 from sunlight.
  Interventions: Other: Precision Bred Vitamin D-rich Tomato Soup
- Soup Made with Wild-Type (Store-bought) Tomatoes (Placebo Comparator): In this soup, store-bought (wild-type) tomatoes contain negligible amounts of 7-DHC and no vitamin D3.
  Interventions: Other: Wild-type (store-bought) Tomato Soup
- Soup Made with Wild-Type (Store-bought) Tomatoes with Vitamin D3 Supplement (Active Comparator): In this soup, store-bought (wild-type) tomatoes are used and supplemented with vitamin D3 (lanolin).
  Interventions: Other: Wild-type (store-bought) Tomato with vitamin D supplementation Soup

INTERVENTIONS:
Other: Precision Bred Provitamin D-rich Tomato Soup — Participants will consume one tomato soup every day for 21 days as part of their normal diet.
  Arms: Soup with Precision Bred Tomatoes (Provitamin D-rich, No UV-Treatment)
Other: Precision Bred Vitamin D-rich Tomato Soup — Participants will consume one tomato soup everyday for 21-days as part of their normal diet.
  Arms: Soup with Precision Bred Tomatoes (Vitamin D-rich, UV-Treated)
Other: Wild-type (store-bought) Tomato Soup — Participants will consume one tomato soup every day for 21 days as part of their normal diet.
  Arms: Soup Made with Wild-Type (Store-bought) Tomatoes
Other: Wild-type (store-bought) Tomato with vitamin D supplementation Soup — Participants will consume one tomato soup everyday for 21 days as part of their normal diet.
  Arms: Soup Made with Wild-Type (Store-bought) Tomatoes with Vitamin D3 Supplement

SUMMARY:
In the UK, vitamin D deficiency occurs frequently especially during the winter months. Vitamin D biofortified tomatoes have been developed using precision breeding technique by researchers at John Innes Centre. Biofortification uses crop breeding to increase the nutritional value of crops. The goal of the ViTaL-D study is to examine whether the vitamin D biofortified tomatoes when eaten as a soup can increase blood levels of vitamin D in men and women with vitamin D deficiency. Additionally, researchers will learn if the tomato soups are feasible and safe to eat everyday. The main questions the study aims to answer are:

* Does vitamin D biofortified tomatoes increase vitamin D levels in men and women with low blood levels of vitamin D?
* Is consuming vitamin D biofortified tomatoes safe and easy to eat everyday as a soup?

Researchers will compare how four types of tomato soup increase blood vitamin D levels. The four types of soup are:

* Soup with vitamin D biofortified tomatoes
* Soup with provitamin D biofortified tomatoes
* Soup with store-bought tomatoes not containing vitamin D
* Soup with store-bought tomatoes with added vitamin D

Participants will:

* Eat one of the four types of tomato soup every day for 21 days.
* Visit the clinic once every 7 days after a 12 hour fast for body measurements, tests, and surveys.
* Keep a daily diary when soups are eaten and when time is spent outside.

DETAILED DESCRIPTION:
The ViTaL-D study is a 21-day randomized, double-blind, placebo-controlled four-arm parallel pilot study conducted at the NIHR (National Institute for Health and Care Research) Norfolk Clinical Research Facility (CRF) in the Quadram Institute in Norwich. Researchers are seeking adult (at least 18 years and older) men and women who have serum 25-hydroxyvitamin D (25[OH]D) levels between 25-40 nmol/L to determine whether soups made with precision bred, biofortified vitamin D tomatoes will increase vitamin D levels. There are a total of 6 study visits (1 consent visit, 1 screening visit, and 4 short visits). At these visits, anthropometric measurements and vital signs will be collected. Participants will be asked to complete questionnaires (food frequency, international physical activity, and sensory evaluation). They will record their daily consumption of soup as well as their daily sun exposure and wear a UV tracker when they are outdoors.

Researchers will measure fasting blood samples for serum 25[OH]D, serum electrolytes, calcium, phosphorous, parathyroid hormone, cholesterol, triglycerides, plasma lycopene, plasma beta carotene, and bone turnover biomarkers. Participants will be given the choice to donate optional samples of saliva and/or 24 hour urine collection. For these optional samples, researchers will quantify vitamin D metabolites (7-DHC, 1,25(OH)2D, 24,25(OH)2D, and C-3 epi 25(OH)D) in saliva and urine as well as vitamin D binding protein in saliva.

Participants will consume one of four soups everyday for 21-days. The four soups are described as such:

* Soup with precision bred tomatoes biofortified with provitamin D (7-dehydrocholesterol-rich, No UV-Treatment). This soup is made with precision bred tomatoes. Tomatoes have been engineered to accumulate 7-dehydrocholesterol (7-DHC, also called provitamin D, a precursor of vitamin D3). The bioefficacy of the provitamin D in the diet is largely unknown.
* Soup with precision bred tomatoes (Vitamin D-rich, UV-Treated) This soup is made with the same precision bred tomatoes, but in this case, the tomatoes have been treated with ultraviolet (UV) light to convert the accumulated 7-DHC into vitamin D3. UV exposure mimics the natural process by which human skin synthesizes vitamin D3 from sunlight.
* Soup with store bought tomatoes (placebo). In this soup, store bought conventional tomatoes contain negligible amounts of 7-DHC and no vitamin D3. This soup is the placebo soup.
* Soup with store bought tomatoes supplemented with Vitamin D3. In this soup, same store-bought tomatoes will be supplemented with vitamin D (from lanolin).

ELIGIBILITY:
Inclusion Criteria:

* Be willing to eat a tomato soup daily for 21 days.
* Have access to a smartphone or tablet device and internet access.
* Be at least 18 years old
* Be able to understand the study and provide informed consent
* Have serum 25-hydroxyvitamin D (25[OH]D) levels between 25-40 nmol/L
* Body Mass Index 18.5 to 35 kg/m2
* Live within 40 miles of the Quadram Institute.

Exclusion Criteria:

* Have a known allergy or intolerance to tomatoes or to any of the soup components (tomatoes, milk, wheat, lanolin are the major allergens, but a detailed list is in Annex 16) of the test soups.
* Currently undergoing treatment or on medications for hypo/hypercalcaemia, hypo/hyperparathyroidism, kidney stones, or bone diseases.
* Have anaemia, immunocompromised or viral infections that may compromise immunity. This will be assessed on a case-by-case basis by QI medical advisor.
* Have any acute or chronic illnesses that affects the outcome of the study such as a gastrointestinal disorder. This will be assessed on a case-by-case basis by Quadram Institute medical advisor.
* Have just started taking or changed dose of vitamin D supplement in the month prior to the start of the intervention or at any point during the intervention, or are regularly taking more than 400 International Units (IU) of vitamin D.
* Are on a routine regimen of vitamin D supplementation over 400 IU who have begun supplementation or had changes in their dose a month prior or have changes during the course of the study.
* Are on any medication regimen that may alter vitamin D absorption they are as follow but not limited to; bile acid sequestrants, hormone replacement therapy, thiazides, calcium channel blockers, isoniazid, anti-seizure medications, and antacids.
* Any dietary restriction that prevents the consumption of the study soups or follow a diet programme which requires fasting for multiple days (soups are not suitable for vegans).
* Have abnormally low or high blood pressure (i.e. ≤90/60, ≥160/100).
* Plan to become pregnant during the study duration, pregnant or breastfeeding.
* Are currently taking part in an intervention study.
* Are a registered blood donor and have donated a large quantity of blood within the last 6 weeks. Registered blood donors should abstain from blood donations for the duration of the study.
* Are unable to give written or verbal informed consent
* Unable to provide your GP contact details.
* Fall under the line management structure or live in the same household with any of the research team, or the QIB Human Studies Team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in plasma lycopene and beta carotene to assess adherence | Day 0 and Day 21
  Fasting plasma total carotenoids and total lycopene
Differences in soup acceptability using sensory evaluation questionnaires as a measure of adherence | Screening visit (Day -60 to -1), Day 1, and Day 21
  Soup acceptability will be measured using a 9-point hedonic scale and 5 point Just-about-Right scale
Assess changes in eating pattern due to daily consumption of soup | Day 0 and Day 21
  VioScreen Food frequency questionnaire
Changes in serum 25-hydroxy vitamin D (25(OH)D) to monitor safety | Day 0 and Day 21
  Fasting serum 25(OH)D levels
Changes in serum electrolytes, calcium and phosphorous to monitor safety | Day 0 and Day 21
  Fasting serum electrolytes, calcium and phosphorus
Change in parathyroid hormone to assess safety | Day 0 and Day 21
  Fasting plasma parathyroid hormone
Assess change in bone turnover biomarkers on serum 25(OH)D levels | Day 0 and Day 21
  Fasting serum procollagen Type 1 N-Terminal Propeptide and Collagen Type 1 Cross-Linked C Telopeptide (P1NP and CTx)
Measure changes in sunlight exposure | Day 0 and Day 21
  Quantify sunlight exposure using Outdoor Skin Assessment, Sun-a-Wear UV tracker UV (duration UV exposure and UV Index)
Measure changes in physical activity | Day 0 and Day 21
  Physical activity will be measured using the International Physical Activity Questionnaire - short version

SECONDARY OUTCOMES:
Treatment effects of daily tomato soup consumption on vitamin D3 or its precursor (7-DHC) on serum 25(OH)D, PTH, cholesterol | Day 21
  Fasting serum 25(OH)D levels Fasting plasma PTH Fasting serum cholesterol, triglycerides, and 25(OH)D levels
Quantify differences in vitamin D metabolites | Day 0 and Day 21
  Vitamin D metabolites measured in serum and urine are provitamin (7-DHC), 1,25(OH)2D, 24,25(OH)2D, and C-3 epi 25(OH)D)
Changes in the quantity of vitamin D and their binding proteins in saliva | Day 0 and Day 21
  Vitamin D metabolites (provitamin (7-DHC), 1,25(OH)2D, 24,25(OH)2D, and C-3 epi 25(OH)D) will be measured in non-stimulated and stimulated saliva Vitamin D binding protein will be measured in non-stimulated and stimulated saliva
Correlate salivary vitamin D and salivary vitamin D binding protein and serum 25(OH)D levels | Day 0 and Day 21
  Vitamin D metabolites (provitamin (7-DHC), 1,25(OH)2D, 24,25(OH)2D, and C-3 epi 25(OH)D) in non-stimulated and stimulated saliva collection Fasting serum 25(OH)D

CONTACTS AND LOCATIONS:
Overall Officials: Martin Warren, PhD, Principal Investigator — Quadram Institute Bioscience
Locations (1):
- Quadram Institute Bioscience, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data which complies with General Data Protection Regulations will be shared